CLINICAL TRIAL: NCT00802737
Title: A Single-arm, International, Multi-center Trial Investigating the Efficacy and Safety of Ofatumumab Retreatment and Maintenance in CLL Patients Who Progressed Following Response or Stable Disease After Ofatumumab Treatment in Hx-CD20-406
Brief Title: Efficacy and Safety of Ofatumumab Retreatment and Maintenance Treatment in Patients With B-cell Chronic Lymphocytic Leukemia (CLL)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Genmab (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 111827; GEN416
Record Dates: First submitted 2008-12-04; First posted 2008-12-05 (Estimated); Results first posted 2012-06-26 (Estimated); Last update posted 2014-05-14 (Estimated); Status verified 2014-04

CONDITIONS: Leukaemia, Lymphocytic, Chronic
Keywords: Maintenance; Retreatment; Chronic lymphocytic leukemia; B-Cell Chronic Lymphocytic Leukemia; Ofatumumab
MeSH Terms: conditions — Leukemia, B-Cell; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — ofatumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ofatumumab (Experimental): Eight once weekly infusions (1 x 300 mg + 7 x 2000 mg), then 2000 mg once monthly for two years
  Interventions: Drug: Ofatumumab

INTERVENTIONS:
Drug: Ofatumumab — Eight once weekly infusions (1 x 300 mg + 7 x 2000 mg), then 2000 mg once monthly for two years
  Other Names: HuMax-CD20

SUMMARY:
The purpose of the trial is to investigate the efficacy and safety of ofatumumab retreatment and maintenance in patients with chronic lymphocytic leukemia who have previously responded or had disease stabilization after ofatumumab in an ongoing trial (Hx-CD20-406).

ELIGIBILITY:
Inclusion Criteria:

* Has responded to ofatumumab treatment (CR, nPR, PR) or has had SD at least up to and including visit number 14 (24 weeks after first infusion) in the Hx-CD20-406 trial.
* Has disease progression after visit number 14 (24 weeks after first infusion) in the Hx CD20 406 trial.
* Received at least eight ofatumumab infusions.
* Has active CLL with an indication for treatment.
* Has Eastern Cooperative Oncology Group (ECOG) performance status grade 0, 1 or 2.
* Provides signed informed consent, following receipt of verbal and written information about the trial, before any trial related activity is carried out.
* If previously treated in GEN416 (this trial), the patient must have achieved CR with subsequent disease progression 24 weeks or later after the first infusion in the GEN416 trial.

Exclusion Criteria:

* The disease has transformed to more aggressive B-cell malignancies (e.g. diffuse large B-cell lymphoma, Richter's syndrome or prolymphocytic leukemia).
* Has a suspected treatment requiring malignancy other than CLL.
* Has received treatment other than ofatumumab within two weeks prior to visit 2.
* Has clinically significant cardiac disease including unstable angina, acute myocardial infarction within six months from visit 1, congestive heart failure (NYHA III IV), and arrhythmia requiring therapy, with the exception of clinically non-significant extra systoles or minor conduction abnormalities.
* Has significant concurrent, uncontrolled medical condition including, but not limited to, renal, hepatic, hematological, gastrointestinal, endocrine, pulmonary, neurological, cerebral or psychiatric disease.
* Has a history of significant cerebrovascular disease.
* Is known HIV positive.
* Has positive serology for hepatitis B, defined as a positive test for HBsAg and/or positive tests for both anti-HBs and anti-HBc.
* Has known or suspected hypersensitivity to components of the IMP.
* Has received treatment with any non-marketed drug substance or experimental therapy other than ofatumumab within four weeks prior to visit 2.
* Currently participates in any other interventional clinical trial other than Hx-CD20-406.
* Known or suspected to not being able to comply with a trial protocol (e.g. due to alcoholism, drug dependency or psychiatric disorder).
* Is breast feeding (women only).
* Has a positive pregnancy test at screening (women only).
* Is not willing to use adequate contraception during the trial and one year after last dose of ofatumumab (women only). Adequate contraception is defined as hormonal birth control or intrauterine device. For patients in the US the use of double barrier method is considered adequate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2009-01; Primary Completion 2011-09 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- Sweden (2):
  - GSK Investigational Site, Örebro
  - GSK Investigational Site, Stockholm

REFERENCES:
- [Derived] van Oers MH, Kuliczkowski K, Smolej L, Petrini M, Offner F, Grosicki S, Levin MD, Gupta I, Phillips J, Williams V, Manson S, Lisby S, Geisler C; PROLONG study investigators. Ofatumumab maintenance versus observation in relapsed chronic lymphocytic leukaemia (PROLONG): an open-label, multicentre, randomised phase 3 study. Lancet Oncol. 2015 Oct;16(13):1370-9. doi: 10.1016/S1470-2045(15)00143-6. Epub 2015 Sep 13. PMID 26377300

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Per study protocol
Pre-assignment Details: Completed study Hx-CD20-406 (Study OMB111773; NCT00349349)
Groups:
- 2000 mg Ofatumumab + DR: Participants (Par.) who had responded to ofatumumab or had stable disease in Hx-CD20-406 (Study OMB111773; NCT00349349) and then progressed were offered retreatment and maintenance. For retreatment, ofatumumab intravenous (iv) infusion was initiated at 300 milligrams (mg), followed by seven weekly 2000 mg infusions. For the maintenance of responders, participants received 24 monthly infusions of 2000 mg for up to 24 months, for a total duration of treatment of up to 26 months after which, if possible, the par. entered the Follow-up phase (Months 29-44). These participants were classified as double refractory (DR), defined as participants who were enrolled in Study Hx-CD20-406 and were refractory to both fludarabine and alemtuzumab. Par. with disease progression entered the Extended Follow-up phase (Months 47 to 62).
- 2000 mg Ofatumumab + BFR: Participants who had responded to ofatumumab or had stable disease in Hx-CD20-406 and then progressed were offered retreatment and maintenance. For retreatment, ofatumumab iv infusion was initiated at 300 mg, followed by seven weekly 2000 mg infusions. For the maintenance of responders, participants received 24 monthly infusions of 2000 mg for up to 24 months, for a total duration of treatment of up to 26 months after which, if possible, the par. entered the Follow-up phase (Months 29-44). These participants were classified as bulky fludarabine refractory (BFR), defined as participants who were enrolled in the study and were refractory to fludarabine with bulky lymphadenopathy. Par. with disease progression entered into the Extended Follow-up phase (Months 47 to 62).
- 2000 mg Ofatumumab + Other: Participants who had responded to ofatumumab or had stable disease in Hx-CD20-406 and then progressed were offered retreatment and maintenance. For retreatment, ofatumumab iv infusion was initiated at 300 mg, followed by seven weekly 2000 mg infusions For the maintenance of responders, participants received 24 monthly infusions of 2000 mg for up to 24 months, for a total duration of treatment of up to 26 months after which, if possible, the par. entered the Follow-up (Months 29-44). These participants were classified as "other," defined as participants who were enrolled in the study but did not meet criteria for DR or BFR. Par. with disease progression entered the Extended Follow-up phase (Months 47 to 62).
Period: Overall Study
Arm/Group | 2000 mg Ofatumumab + DR | 2000 mg Ofatumumab + BFR | 2000 mg Ofatumumab + Other
Started | 17 | 11 | 1
Completed | 0 | 0 | 0
Not Completed | 17 | 11 | 1
Not completed — Withdrawn due to Disease Progression | 9 | 3 | 0
Not completed — Death | 6 | 5 | 1
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Received Prohibited Therapy | 1 | 0 | 0
Not completed — Ongoing CLL-Treatment | 0 | 1 | 0
Not completed — Participant too Unwell | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 2000 mg Ofatumumab + DR | 2000 mg Ofatumumab + BFR | 2000 mg Ofatumumab + Other | Total
Number analyzed (Participants) | 17 | 11 | 1 | 29
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.8 (5.83) | 66.9 (9.08) | 84.0 (NA) — A standard deviation of the mean was not calculated for one participant. | 66.3 (7.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 1 | 9
  Male | 13 | 7 | 0 | 20
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 1 | 0 | 0 | 1
  White | 16 | 11 | 1 | 28

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants (Par.) Classified as Responders (Rs) and Non-responders (NRs) for Objective Response in Accordance With the National Cancer Institute Working Group (NCIWG) 1996 Guidelines
Description: Par. with complete remission (CR), nodular partial remission (nPR), and partial remission (PR) on 2 consecutive visits >=56 days apart were classified as Rs; those with stable disease (SD)/progressive disease (PD) were classified as NRs. Per the NCIWG 1996 guidelines: CR; no lymphadenopathy/hepatomegaly/splenomegaly/constitutional symptoms, normal hematology, normocellular bone marrow sample for age, <30% lymphocytes (LC), no lymphoid nodule; PR: >=50% decrease in LC/lymphadenopathy; nPR: persistent bone marrow nodules; PD: new lesion or increase by >=50% from baseline; SD: no CR, PR, or PD.
Time Frame: Start of treatment (Week 0/Visit 2) until Week 52
Population: Full Analysis Set (FAS): all participants who had been exposed to study drug irrespective of their compliance to the planned course of treatment. Some participants were not evaluable (NE) due to participant withdraw, refusal, non-trial drug-related adverse events, and death.
Measure: Number; unit: participants
Arm/Group | 2000 mg Ofatumumab + DR | 2000 mg Ofatumumab + BFR | 2000 mg Ofatumumab + Other
Number analyzed (Participants) | 17 | 11 | 1
participants
  Responders with CR | 2 | 0 | 0
  Responders with nPR | 0 | 0 | 0
  Responders with PR | 2 | 2 | 1
  Non-responders with SD | 8 | 7 | 0
  Non-responders with PD | 3 | 0 | 0
  NE | 2 | 2 | 0
Statistical Analysis 1: Comparison: 2000 mg Ofatumumab + DR; Test type: Superiority or Other; proportion of responders = 0.24, 95% CI 2-sided [0.07 to 0.50] — Two-sided 95% exact confidence intervals were calculated based on the binomial distribution. The estimated value was calculated using the number of responders (CR+nPR+PR) as the numerator and the total number of par. in the group as the denominator
Statistical Analysis 2: Comparison: 2000 mg Ofatumumab + BFR; Test type: Superiority or Other; proportion of responders = 0.18, 95% CI 2-sided [0.02 to 0.52] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: 2000 mg Ofatumumab + Other; Test type: Superiority or Other; proportion of responders = 1.00, 95% CI 2-sided [0.03 to 1.00] — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Duration of Response
Description: Duration of response is defined as the time from the initial response (first visit at which response is observed) to progression or death. If the participant had progression between scheduled visits, no progression at the end of the trial, treatment discontinuation for undocumented progression, treatment discontinuation for toxicity or other reason, new anti-cancer treatment, and experienced death or progression after two or more missed visits in a row the endpoint was censored.
Time Frame: From the time of the initial response until progression or death (average of 14.1 study months)
Population: FAS
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | 2000 mg Ofatumumab + DR | 2000 mg Ofatumumab + BFR | 2000 mg Ofatumumab + Other
Number analyzed (Participants) | 17 | 11 | 1
months | NA [7.2 to NA] — There were not enough events on the survival curve to estimate a median or upper limit of confidence interval. | NA [24.1 to NA] — There were not enough events on the survival curve to estimate a median or upper limit of confidence interval | NA [NA to NA] — There were not enough events on the survival curve to estimate a median or confidence interval.

3. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS is defined as the time from randomization until progression (prog.)/death. Prog. events are defined by well-documented and verifiable data; other data are censored. If the par. had prog. between scheduled visits, died before the first assessment, or died between adequate visits, the endpoint was considered progressed. If there was no prog. at the end of the trial, treatment discontinuation for undocumented prog./toxicity/other reason, new anti-cancer treatment, and death/prog. after >=2 missed visits in a row, the endpoint was censored. Clinical prog. is not considered as a prog. endpoint.
Time Frame: Start of treatment (Week 0 of Visit 2) until progression or death (average of 14.1 study months)
Population: FAS
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | 2000 mg Ofatumumab + DR | 2000 mg Ofatumumab + BFR | 2000 mg Ofatumumab + Other
Number analyzed (Participants) | 17 | 11 | 1
months | 7.9 [3.2 to 12.9] | 7.2 [2.0 to 11.6] | NA [NA to NA] — There were not enough events on the survival curve to estimate a median or confidence interval.

4. Secondary Outcome: Time to Next Chronic Lymphocytic Leukemia (CLL) Treatment
Description: Time to next chronic lymphocytic leukemia (CLL) treatment is defined as the time from treatment allocation/randomization (Visit 2) until the time of the first administration of the next CLL treatment other than ofatumumab (or HuMaxCD20, a fully human monoclonal antibody to CD20 that is expressed on the surface of B-cells).
Time Frame: Time from start of study treatment (Week 0 of Visit 2) until the time of first administration of a CLL treatment other than ofatumumab (average of 14.8 study months)
Population: FAS
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | 2000 mg Ofatumumab + DR | 2000 mg Ofatumumab + BFR | 2000 mg Ofatumumab + Other
Number analyzed (Participants) | 17 | 11 | 1
months | 13.9 [3.9 to NA] — There were not enough events on the survival curve to estimate the upper limit of the confidence interval. | 11.6 [7.0 to NA] — There were not enough events on the survival curve to estimate the upper limit of the confidence interval. | NA [NA to NA] — There were not enough events on the survival curve to estimate a median or confidence interval.

5. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from allocation to death.
Time Frame: Time from start of study treatment (Week 0 of Visit 2) until date of death or time that participant was no longer followed (median of 18.0 months)
Population: FAS
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | 2000 mg Ofatumumab + DR | 2000 mg Ofatumumab + BFR | 2000 mg Ofatumumab + Other
Number analyzed (Participants) | 17 | 11 | 1
months | 27.6 [5.4 to NA] — There were not enough events on the survival curve to estimate the upper limit of the confidence interval. | 11.3 [5.3 to NA] — There were not enough events on the survival curve to estimate the upper limit of the confidence interval. | 12.3 [NA to NA] — There were not enough events on the survival curve to estimate a confidence interval.

6. Secondary Outcome: Median Percent Change of Tumor Size (Sum of Products Dimensions [SPD]) From Baseline (Visit 2) at Month 4
Description: Reduction in tumor size was measured as the percent change in the sum of the products of the diameters of the largest abnormal lymph nodes from Baseline to Week 24. Percent change was calculated as (Week 24 SPD minus Baseline SPD)/Baseline SPD * 100.
Time Frame: Baseline (Visit 2) and Month 4
Population: FAS. Measurement of tumor size was completed by physical examination for participants remaining in the study at Month 4. Only participants with a baseline value and a post-baseline value at Month 4 were included in the calculation.
Measure: Median (Full Range); unit: Percent change in tumor size
Arm/Group | 2000 mg Ofatumumab + DR | 2000 mg Ofatumumab + BFR | 2000 mg Ofatumumab + Other
Number analyzed (Participants) | 8 | 6 | 1
Percent change in tumor size | -55.3 [-100 to 157] | -64.8 [-82 to 3] | 0 [0 to 0]

7. Secondary Outcome: Median Percent Change of Tumor Size (Sum of Products Dimensions [SPD]) From Baseline (Visit 2) at Month 12
Description: Reduction in tumor size was measured by the percentage change in the sum of products of the diameters of the largest abnormal lymph nodes from Baseline to Month 12. Percent change was calculated as (Month 12 SPD minus Baseline SPD)/Baseline SPD * 100.
Time Frame: Baseline (Visit 2) and Month 12
Population: FAS. No participants in the 2000 mg Ofatumumab + Other treatment arm were able to contribute to this measure. Measurement of tumor size was completed by physical examination for participants remaining in the study at Month 12. Only participants with a baseline value and a post-baseline value at Month 12 were included in the calculation.
Measure: Median (Full Range); unit: Percent change in tumor size
Arm/Group | 2000 mg Ofatumumab + DR | 2000 mg Ofatumumab + BFR | 2000 mg Ofatumumab + Other
Number analyzed (Participants) | 4 | 1 | 0
Percent change in tumor size | -65.2 [-100 to 0] | -68.9 [-68.9 to -68.9] |

8. Secondary Outcome: Median Percent Change of Tumor Size (Sum of Products Dimensions [SPD]) From Baseline (Visit 2) at Month 24
Description: Reduction in tumor size was measured by the percentage change in the sum of products of the diameters of the largest abnormal lymph nodes from Baseline to Month 24. Percent change was calculated as (Month 24 SPD minus Baseline SPD)/Baseline SPD * 100.
Time Frame: Baseline (Visit 2) and Month 24
Population: FAS. No participants in the 2000 mg Ofatumumab + Other treatment arm were able to contribute to this measure. Measurement of tumor size was completed by physical examination for participants remaining in the study at Month 24. Only participants with a baseline value and a post-baseline value at Month 24 were included in the calculation.
Measure: Median (Full Range); unit: Percent change in tumor size
Arm/Group | 2000 mg Ofatumumab + DR | 2000 mg Ofatumumab + BFR | 2000 mg Ofatumumab + Other
Number analyzed (Participants) | 2 | 1 | 0
Percent change in tumor size | -83.3 [-100 to -67] | -64.0 [-64 to -64] |

9. Secondary Outcome: Number of Participants With Negative and Positive Human Anti-human Antibody (HAHA) Results at the Time of Screening and Post Ofatumumab
Description: HAHAs are indicators of immunogenicity to ofatumumab. HAHA levels were assessed for each participant at the end of participation in the study (at their last visit). A positive HAHA status indicates a positive enzyme-linked immunosorbent assay (ELISA) result, an inconclusive status indicates a negative ELISA result at ofatumumab concentration above the threshold at which ofatumumab may interfere with the assay, and a negative status indicates a negative ELISA result at ofatumumab concentration below the threshold.
Time Frame: Screening and post ofatumumab (up to Study Month 32)
Population: FAS. During the study, samples were to be taken at the last visit; however, this may not have been possible, such as in cases of death, or when the visit was not obvious as the "last visit." Therefore, some samples were not available or were not collected.
Measure: Number; unit: participants
Groups:
- Total: This arm includes a total of all three arms combined.
Arm/Group | 2000 mg Ofatumumab + DR | 2000 mg Ofatumumab + BFR | 2000 mg Ofatumumab + Other | Total
Number analyzed (Participants) | 17 | 11 | 1 | 29
participants
  Screening, Positive, n=15 , 11, 1, 27 | 0 | 0 | 0 | 0
  Screening, Inconclusive, n = 15 , 11 , 1, 27 | 5 | 6 | 0 | 11
  Screening, Negative, n = 15 , 11 , 1, 27 | 10 | 5 | 1 | 16
  Post-ofatumumab, Positive, n = 12 , 8 , 1, 21 | 0 | 0 | 0 | 0
  Post-ofatumumab, Inconclusive, n=12 , 8, 1, 21 | 9 | 8 | 1 | 18
  Post-ofatumumab, Negative, n =12 , 8, 1 , 21 | 3 | 0 | 0 | 3

10. Secondary Outcome: Number of Participants Who Experienced Any Adverse Event
Description: An adverse event (AE) is defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which did not necessarily have a causal relationship with the treatment. A list of AEs experienced in the study with a frequency threshold of 5% can be found in the AE section of this results record.
Time Frame: From the first infusion (Visit 2/Week 0) until the last visit of the Extended Follow-up Phase (up to Study Month 26 [visit 34])
Population: FAS
Measure: Number; unit: participants
Arm/Group | 2000 mg Ofatumumab + DR | 2000 mg Ofatumumab + BFR | 2000 mg Ofatumumab + Other
Number analyzed (Participants) | 17 | 11 | 1
participants | 15 | 11 | 1

11. Secondary Outcome: Number of Participants With the Indicated Major Infections
Description: The data collected for this analysis are reported in the overall Serious Adverse Events (SAEs) of infections rather than reported separately for this specific analysis. This is a conservative approach for reporting all infectious SAEs in order to ensure that all of the infectious SAEs are represented.
Time Frame: as for outcome 10
Population: FAS
Arm/Group | 2000 mg Ofatumumab + DR | 2000 mg Ofatumumab + BFR | 2000 mg Ofatumumab + Other
Number analyzed (Participants) | 0 | 0 | 0

12. Secondary Outcome: Number of Participants With Infections Requiring Hospitalization or Intravenous Antibiotics
Description: The data collected for this analysis are reported in the overall SAEs of infections rather than reported separately for this specific analysis. This is a conservative approach for reporting all infectious SAEs in order to ensure that all of the infectious SAEs are represented.
Time Frame: as for outcome 10
Population: FAS
Arm/Group | 2000 mg Ofatumumab + DR | 2000 mg Ofatumumab + BFR | 2000 mg Ofatumumab + Other
Number analyzed (Participants) | 0 | 0 | 0

13. Secondary Outcome: Cmax and Ctrough at Visit 2 (Week 0) and at Visit 14 (Month 4)
Description: Cmax is defined as the maximum concentration of drug in plasma samples (collected at the end of the infusion). Ctrough is defined as the concentration of drug in plasma samples at the end of a dosing interval (collected directly before next administration). Ctrough before the first infusion represents residual ofatumumab from participation in Study Hx-CD20-406.
Time Frame: Visit 2 (Week 0) and Visit 14 (Month 4)
Population: FAS. Data are provided for the number of participants attending each visit. Participants withdrawn during the study were not analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: Milligrams per liter (mg/L)
Arm/Group | 2000 mg Ofatumumab + DR | 2000 mg Ofatumumab + BFR | 2000 mg Ofatumumab + Other | Total
Number analyzed (Participants) | 17 | 11 | 1 | 29
Milligrams per liter (mg/L)
  Cmax Visit 2, n= 16, 11, 1, 28 | 54.8 [30.7 to 97.7] | 58.8 [38.6 to 89.5] | 110 [NA to NA] — The 95% CI could not be calculated due to the sample size (n=1). | 57.7 [40.7 to 82.0]
  Cmax Visit 14, n= 8, 5, 0, 13 | 617 [413 to 922] | 708 [352 to 1424] | NA [NA to NA] — Participants in group Ofatumumab + Other did not have a sample collection at Visit 14. | 651 [482 to 877]
  Ctrough Visit 2, n= 16, 11, 1, 28 | 1.1 [0.32 to 4.0] | 2.8 [1.1 to 7.5] | 0.0 [NA to NA] — The 95% CI could not be calculated due to the sample size (n=1). | 1.7 [0.77 to 3.6]
  Ctrough Visit 14, n= 8, 5, 0, 13 | 42.6 [6.4 to 285] | 59.5 [4.7 to 757] | NA [NA to NA] — Participants in group Ofatumumab + Other did not have a sample collection at Visit 14. | 48.5 [13.6 to 173]

ADVERSE EVENTS:
Time Frame: On-treatment serious adverse events (SAEs) and non-serious adverse events (AEs) were collected from the first dose of investigational product until the last visit of the Extended Follow-up Phase (up to Study Month 26 [visit 34]).
Description: SAEs and non-serious AEs were reported for members of the Safety Population, comprised of all participants randomized to treatment who received >=1 dose of trial medication.
Arm/Group | 2000 mg Ofatumumab + DR | 2000 mg Ofatumumab + BFR | 2000 mg Ofatumumab + Other
Serious Adverse Events (participants affected / at risk) | 11/17 | 10/11 | 1/1
Other Adverse Events (participants affected / at risk) | 15/17 | 11/11 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 2000 mg Ofatumumab + DR (N=17) | 2000 mg Ofatumumab + BFR (N=11) | 2000 mg Ofatumumab + Other (N=1)
Bronchopneumonia (Infections and infestations) | 2 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 2 | 0
Candida pneumonia (Infections and infestations) | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 1 | 0
Infection (Infections and infestations) | 1 | 0 | 0
Lung infection pseudomonal (Infections and infestations) | 0 | 1 | 0
Pneumocystis jiroveci pneumonia (Infections and infestations) | 0 | 1 | 0
Rhinitis (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 3 | 0 | 0
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0
Disease progression (General disorders) | 2 | 1 | 1
Pyrexia (General disorders) | 1 | 1 | 0
Death (General disorders) | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0
Chronic lympocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Chronic lymphocytic leukaemia refractory (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Melanoma, recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Malignant neoplasm of pleura (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Enteritis (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 1 | 0
Weight decreased (Investigations) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Femoral artery occlusion (Vascular disorders) | 1 | 0 | 0
Infection Respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Respiratory tract infection fungal (Infections and infestations) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 2000 mg Ofatumumab + DR (N=17) | 2000 mg Ofatumumab + BFR (N=11) | 2000 mg Ofatumumab + Other (N=1)
Diarrhea (Gastrointestinal disorders) | 4 | 5 | 1
Nausea (Gastrointestinal disorders) | 5 | 2 | 0
Vomiting (Gastrointestinal disorders) | 4 | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 4 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 3 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 2 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 1 | 0
Gingivitis (Gastrointestinal disorders) | 0 | 2 | 0
Paraesthesia oral (Gastrointestinal disorders) | 1 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0
Hiatus hernia (Gastrointestinal disorders) | 1 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 1 | 0
Oral pain (Gastrointestinal disorders) | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0
Tongue blistering (Gastrointestinal disorders) | 0 | 1 | 0
Bronchitis (Infections and infestations) | 2 | 1 | 0
Furuncle (Infections and infestations) | 1 | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0 | 1
Infected bites (Infections and infestations) | 2 | 0 | 0
Respiratory tract infection (Infections and infestations) | 1 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 0
Candidiasis (Infections and infestations) | 0 | 1 | 0
Erysipelas (Infections and infestations) | 1 | 0 | 0
Fungal infection (Infections and infestations) | 0 | 1 | 0
Fungal skin infection (Infections and infestations) | 1 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Lung infection (Infections and infestations) | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 1 | 0
Rhinitis (Infections and infestations) | 1 | 0 | 0
Skin infection (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0
Chills (General disorders) | 1 | 4 | 1
Pyrexia (General disorders) | 4 | 3 | 0
Oedema peripheral (General disorders) | 1 | 3 | 0
Chest pain (General disorders) | 2 | 0 | 0
Fatigue (General disorders) | 0 | 2 | 0
Infusion site extravasation (General disorders) | 0 | 2 | 0
Asthenia (General disorders) | 0 | 1 | 0
Chest discomfort (General disorders) | 0 | 1 | 0
Influenza like illness (General disorders) | 0 | 1 | 0
Oedema (General disorders) | 1 | 0 | 0
Back pains (Musculoskeletal and connective tissue disorders) | 3 | 3 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Musculoskeletal chest pains (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 4 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 2 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 2 | 0
Cachexia (Metabolism and nutrition disorders) | 0 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Magnesium deficiency (Metabolism and nutrition disorders) | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 3 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 1 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Flushing (Vascular disorders) | 3 | 1 | 0
Hypotension (Vascular disorders) | 1 | 2 | 0
Hypertension (Vascular disorders) | 1 | 1 | 0
Hot flush (Vascular disorders) | 0 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 2 | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Splenomegaly (Blood and lymphatic system disorders) | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 2 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 0
Dizziness postural (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Wound (Injury, poisoning and procedural complications) | 1 | 0 | 0
C-Reactive protein increased (Investigations) | 1 | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0
Platelet count decreased (Investigations) | 0 | 1 | 0
Reticulocyte count increased (Investigations) | 1 | 0 | 0
Weight decreased (Investigations) | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 2 | 0 | 0
Allergy to arthropod bite (Immune system disorders) | 1 | 0 | 0
Conjunctivitis (Eye disorders) | 0 | 1 | 1
Eyelid oedema (Eye disorders) | 0 | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 1 | 0 | 0
Renal impairment (Renal and urinary disorders) | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0
Haemophilus infection (Infections and infestations) | 1 | 0 | 0
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.